CLINICAL TRIAL: NCT03647072
Title: Comparative Clinical and Biochemical Study Evaluating the Effect of Proton Pump I Nhibitors Versus Histamine 2 Receptor Antagonists as an Adjuvant With Chemotherapy in Patients With Non-hodgkin Lymphoma.
Brief Title: PPI Versus Histamine Antagnists as Adjuvant to Chemotherapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, PhDTropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: eman elberry
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — CHOP protocol; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHOP (Active Comparator): CHOP only
  Interventions: Drug: CHOP
- CHOP Plus Lanzoprazole (Active Comparator): CHOP Plus Lanzoprazole 60 mg
  Interventions: Drug: CHOP Plus Lanzoprazole
- CHOP Plus Famotidine (Active Comparator): CHOP Plus Famotidine 40 mg
  Interventions: Drug: CHOP Plus Famotidine

INTERVENTIONS:
Drug: CHOP — CHOP only
  Other Names: CHOP protocol
  Arms: CHOP
Drug: CHOP Plus Lanzoprazole — CHOP plus Lanzoprazole 60 mg
  Other Names: CHOP Plus Lanzoprazole 60
  Arms: CHOP Plus Lanzoprazole
Drug: CHOP Plus Famotidine — CHOP Plus Famotidine 40 mg
  Other Names: CHOP Plus Famotidine 40
  Arms: CHOP Plus Famotidine

SUMMARY:
The study is a Comparative Clinical and Biochemical Study Evaluating the effect of Proton Pump I nhibitors versus histamine 2 Receptor antagonists as an adjuvant with chemotherapy in patients with Non-hodgkin Lymphoma.

DETAILED DESCRIPTION:
The study is a Comparative Clinical and Biochemical Study Evaluating the effect of Proton Pump Inhibitors versus histamine 2 Receptor antagonists as an adjuvant with chemotherapy in patients with Non-hodgkin Lymphoma to compare the difference in efficacy.

ELIGIBILITY:
Inclusion Criteria:

* DLBCL Lymphoma subtype --No comorbid disease

Exclusion Criteria:

* Pregnancy
* Peptic ulcer
* Severe cardiac disease
* Osteoporosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients eith radiological and clinical improvement | 6 months
  Number of patients eith radiological and clinical improvement after cycles of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Sahar K Hegazy, Prof, Principal Investigator — Clinical pharmacy Department- Tanta University; Sahar M El-Haggar, prof, Study Director — Clinical pharmacy Department- Tanta University; Suzan A Alhassanin, Ph D, Study Director — Clinical Oncology Department-Menoufia University; Eman I A El berri, Msc, Principal Investigator — Clinical pharmacy Department-Tanta University
Locations (1):
- Sherief Abd-Elsalam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hegazy SK, El-Haggar SM, Alhassanin SA, El-Berri EI. Comparative randomized trial evaluating the effect of proton pump inhibitor versus histamine 2 receptor antagonist as an adjuvant therapy in diffuse large B-cell lymphoma. Med Oncol. 2021 Jan 4;38(1):4. doi: 10.1007/s12032-020-01452-z. PMID 33394214